CLINICAL TRIAL: NCT03064490
Title: Pembrolizumab, Radiotherapy, and Chemotherapy in Neoadjuvant Treatment of Malignant Esophago-gastric Diseases (PROCEED)
Acronym: PROCEED
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00081010
Record Dates: First submitted 2017-02-22; First posted 2017-02-27 (Actual); Results first posted 2024-03-13 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Locally Advanced Esophageal and Gastric Cancers (EGC)
MeSH Terms: conditions — Stomach Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single arm interventional study (Other): Single arm, non randomized, open label study. Subjects will receive three doses of neoadjuvant pembrolizumab (200 mg administered as an intravenous infusion over 30 minutes every 3 weeks). Pembrolizumab will be administered with weekly standard of care Carboplatin/Paclitaxel concurrent chemo-radiation therapy in the neo-adjuvant setting. Postoperatively, three additional cycles of pembrolizumab (200 mg every 3 weeks) will be administered as adjuvant therapy.
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — Neoadjuvant Pembrolizumab ( 3 cycles) administered concurrently with weekly Carboplatin and Paclitaxel and daily radiation therapy; followed by surgical resection and adjuvant Pembrolizumab ( 3 cycles)
  Other Names: Keytruda

SUMMARY:
This is a single-institution, prospective phase II trial with an initial safety run-in to evaluate the efficacy and safety of neoadjuvant pembrolizumab combined with chemoradiotherapy and adjuvant pembrolizumab in patients with locally advanced esophageal and gastric cancers (EGC). Chemoradiation therapy (45Gy in 25 fractions with concurrent, weekly carboplatin [AUC 2] and paclitaxel [50mg/m2 of BSA]) with three cycles of pembrolizumab will be administered as neoadjuvant therapy. These patients will also receive three cycles of adjuvant pembrolizumab after surgical resection

DETAILED DESCRIPTION:
Enrolled patients will receive three doses of neoadjuvant pembrolizumab (200 mg administered as an intravenous infusion over 30 minutes every 3 weeks). The first dose of pembrolizumab will be administered approximately 14 days prior to initiating radiotherapy. The second dose will be administered three weeks later (week 1 of chemoradiation). The third dose will be administered 3 weeks later (week 4 of chemoradiotherapy). Pembrolizumab will be given every 3 weeks and may be given at the same time as systemic therapy. All patients will receive radiation treatment (45Gy in 25 fractions at 1.8 Gy/fraction) using image-guided radiation therapy with concurrent, weekly carboplatin (AUC 2) and paclitaxel (50mg/m2 of BSA). Restaging will be performed per standard of care approximately 4-8 weeks after completing chemoradiotherapy. Resection will be performed approximately 6-12 weeks after completing chemoradiotherapy per standard of care. Postoperatively, three additional cycles of pembrolizumab (200 mg every 3 weeks) will be administered as adjuvant therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent for the trial.
2. Be 18 years of age or older on day of signing informed consent.
3. Has a pathologic diagnosis of invasive esophageal, gastroesophageal or gastric adenocarcinoma.
4. Staging CT CAP or PET/CT shows no evidence of metastatic disease.
5. Have a performance status of 0-2 on the ECOG Performance Scale.
6. Plan for neoadjuvant chemoradiation.
7. Demonstrate adequate organ function as defined in the study protocol, all screening labs should be performed within 14 days of treatment initiation.
8. Female subject of childbearing potential should have a negative serum pregnancy within 48 hours prior to receiving the first dose of study medication.
9. Female and male subjects of childbearing potential must be willing to use an adequate method of contraception as outlined in the Duke Contraception Policy.

Exclusion Criteria:

1. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
2. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
3. Has a known history of active TB (Bacillus Tuberculosis)
4. Hypersensitivity to pembrolizumab or any of its excipients.
5. Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
6. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy for the current diagnosis of EGC.
7. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer. (all patients with prior radiotherapy must be reviewed by the PI to determine if patient is eligible).
8. Has known metastatic disease. Staging CT C/A/P or PET/CT will be mandatory no more than 45 days prior to enrollment to evaluate for the presence of metastatic disease.
9. Has unresectable disease or is medically inoperable.
10. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with chronic use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
11. Has known history of, or any evidence of active, non-infectious pneumonitis.
12. Has an active infection requiring systemic therapy.
13. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
14. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
15. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
16. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
17. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
18. Has known, active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
19. Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.
20. Has a diagnosis of scleroderma.
21. Has a known history of allogenic stem cell transplant
22. Has received a solid organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2017-10-17 (Actual); Primary Completion 2023-02-24 (Actual); Study Completion 2023-11-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manisha Palta, MD, Principal Investigator — Duke University
Locations (1):
- Duke Cancer Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single Arm Interventional Study
Started | 35
Completed | 30
Not Completed | 5
Not completed — Physician Decision | 5

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm Interventional Study
Number analyzed (Participants) | 35
Age, Continuous [Median (Full Range); unit: years] | 60 [33 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 35
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 33
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Pathologic Complete Response (pCR)
Description: A two-stage design will be used to test the null hypothesis that the true pCR rate is ≤ 0.30 against the alternative hypothesis that the true pCR rate is ≥ 0.50. This design will allow the trial to stop early to accept the null hypothesis. If there are no more than 4 responders (27%) in the first 15 evaluable patients, the trial will stop to accept the null. Otherwise, an additional 15 evaluable patients will be accrued.
Time Frame: up to 20 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm Interventional Study
Number analyzed (Participants) | 30
Participants | 11

2. Secondary Outcome: Safety of the Combined Drug Therapy With Radiation Therapy
Description: The number of Grade 3+ non-hematological adverse events of special interest that occurred will be reported.
Time Frame: Neoadjuvant: from the start of neoadjuvant therapy until surgery, approximately 20 weeks Postoperative: within 30 days after surgery Adjuvant: from the start of adjuvant therapy until 90 days after the last dose of adjuvant therapy
Measure: Number; unit: events
Arm/Group | Single Arm Interventional Study
Number analyzed (Participants) | 34
events
  Rash | 6
  Esophagitis | 2
  Lung infection | 2
  Dyspnea | 1
  Pneumonitis | 3
  Esophageal pain | 2
  Thrombolytic event | 3
  Hyponatremia | 6
  Fever | 4
  Aspartate aminotransferase increased | 2
  Blood bilirubin increased | 1
  Diarrhea | 2
  Colitis | 2
  Dehydration | 2
  Vasovagal reaction | 1
  Syncope | 1
  Glucose intolerance | 1
  Fatigue | 2
  Infection | 1
  Sinus tachycardia | 1
  Hypoxia | 1
  Fall | 1
  Weight loss | 1
  Investigation, other | 1
  GI disorder, other | 1

ADVERSE EVENTS:
Time Frame: Neoadjuvant: from the start of neoadjuvant therapy until surgery, approximately 20 weeks Postoperative: within 30 days after surgery Adjuvant: from the start of adjuvant therapy until 90 days after the last dose of adjuvant therapy
Description: Serious adverse events are defined as Grade 3+ adverse events leading to hospitalization
Arm/Group | Single Arm Interventional Study
All-Cause Mortality (participants affected / at risk) | 9/35
Serious Adverse Events (participants affected / at risk) | 15/35
Other Adverse Events (participants affected / at risk) | 33/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm Interventional Study (N=35)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Gastric anastomotic leak (Injury, poisoning and procedural complications) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 2 (2)
Esophageal anastomotic leak (Injury, poisoning and procedural complications) | 2 (2)
Esophagitis (Gastrointestinal disorders) | 2 (2)
Fever (General disorders) | 3 (4)
Autoimmune disorder (Immune system disorders) | 1 (1)
Lung Infection (Infections and infestations) | 2 (2)
Sepsis (Infections and infestations) | 2 (2)
Wound infection (Infections and infestations) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 6 (6)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural infection (Infections and infestations) | 1 (1)
Thromboembolic event (Vascular disorders) | 3 (3)
Hypotension (Vascular disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 2 (2)
Upper respiratory infection (Infections and infestations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Neutrophil count decreased (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 2 (2) — Fever, treated with IV antibiotics; COVID Positive
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Investigations - Other, specify (Investigations) | 1 (1) — Leukocytosis
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1 (1) — Failure to thrive
Lethargy (Nervous system disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1) — Left ICA terminus aneurysm
Rash (Skin and subcutaneous tissue disorders) | 6 (6)
Esophageal pain (Gastrointestinal disorders) | 2 (2)
Vasovagal reaction (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Glucose intolerance (Metabolism and nutrition disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
Infection (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Weight loss (Investigations) | 1 (1)
Investigations, other (Investigations) | 1 (1)
GI disorder, other (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm Interventional Study (N=35)
Anemia (Blood and lymphatic system disorders) | 33 (51)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 3 (3)
Chest pain - cardiac (Cardiac disorders) | 3 (3)
Sinus tachycardia (Cardiac disorders) | 2 (2)
Endocrine disorders - Other, specify (Endocrine disorders) | 3 (3) — Thyroid Stimulating-Hormone (TSH) descreased; cortisol level decreased; low ACTH; TSH decreased
Hyperthyroidism (Endocrine disorders) | 2 (2)
Hypothyroidism (Endocrine disorders) | 8 (9)
Abdominal pain (Gastrointestinal disorders) | 12 (14)
Bloating (Gastrointestinal disorders) | 3 (4)
Constipation (Gastrointestinal disorders) | 25 (30)
Diarrhea (Gastrointestinal disorders) | 16 (27)
Dyspepsia (Gastrointestinal disorders) | 6 (6)
Dysphagia (Gastrointestinal disorders) | 7 (9)
Esophageal pain (Gastrointestinal disorders) | 7 (11)
Esophagitis (Gastrointestinal disorders) | 29 (41)
Flatulence (Gastrointestinal disorders) | 2 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 4 (5)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 5 (7) — Hematemesis; scant hemoptysis; belching; hematochezia; gas in esophagus creating chest pressure; hematemesis (vomiting bright red blood)
Gastroparesis (Gastrointestinal disorders) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 29 (50)
Oral pain (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 20 (31)
Chills (General disorders) | 6 (6)
Edema limbs (General disorders) | 3 (3)
Fatigue (General disorders) | 33 (53)
Fever (General disorders) | 9 (17)
General disorders and administration site conditions - Other, specify (General disorders) | 4 (4) — Night sweats; weakness; chest tightness
Infusion related reaction (General disorders) | 5 (6)
Pain (General disorders) | 9 (12)
Allergic reaction (Immune system disorders) | 10 (10)
Bronchial infection (Infections and infestations) | 3 (3)
Infections and infestations - Other, specify (Infections and infestations) | 5 (5) — Clostridium Difficile; Lft nostril infection; Atypical pneumonia; aspiration pneumonia
Lung infection (Infections and infestations) | 3 (3)
Phlebitis infective (Infections and infestations) | 3 (3)
Rash pustular (Infections and infestations) | 2 (2)
Skin infection (Infections and infestations) | 3 (3)
Urinary tract infection (Infections and infestations) | 4 (5)
Dermatitis radiation (Injury, poisoning and procedural complications) | 5 (5)
Aspartate aminotransferase increased (Investigations) | 6 (13)
Lymphocyte count decreased (Investigations) | 2 (2)
Neutrophil count decreased (Investigations) | 19 (31)
Platelet count decreased (Investigations) | 24 (43)
White blood cell decreased (Investigations) | 24 (49)
Blood and lymphatic system disorders - Other, specify (Investigations) | 3 (3) — Elevated white blood cell count (2), Elevated neutrophil count (1)
Alanine aminotransferase increased (Investigations) | 8 (13)
Alkaline phosphatase increased (Investigations) | 7 (8)
Blood bilirubin increased (Investigations) | 5 (8)
Creatinine increased (Investigations) | 4 (4)
Investigations - Other, specify (Investigations) | 4 (4) — Elevated white blood cell count; White blood cell/Neutrophil count increased; immunotherapy-related hepatitis
Weight loss (Investigations) | 20 (27)
Anorexia (Metabolism and nutrition disorders) | 10 (10)
Dehydration (Metabolism and nutrition disorders) | 19 (54)
Hyperkalemia (Metabolism and nutrition disorders) | 4 (4)
Hypoalbuminemia (Metabolism and nutrition disorders) | 20 (29)
Hypocalcemia (Metabolism and nutrition disorders) | 5 (5)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (3)
Hypokalemia (Metabolism and nutrition disorders) | 11 (18)
Hypomagnesemia (Metabolism and nutrition disorders) | 6 (7)
Hyponatremia (Metabolism and nutrition disorders) | 27 (58)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 3 (3) — Low protein; Low Uric acid;
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (5)
Dizziness (Nervous system disorders) | 13 (14)
Dysgeusia (Nervous system disorders) | 3 (5)
Headache (Nervous system disorders) | 7 (9)
Nervous system disorders - Other, specify (Nervous system disorders) | 3 (3) — Numbness thumb/pinkie finger Rt finger; Altered sensation noticed on the right posterior 2-3 inches above the knee approximately; jitteriness
Paresthesia (Nervous system disorders) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (4)
Hematuria (Renal and urinary disorders) | 2 (2)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 4 (5) — Urobilinogen elevated; Elevated BUN and BUN/Crea ratio; weak urine stream
Urinary tract pain (Renal and urinary disorders) | 2 (2)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 22 (33)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 11 (18)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 (9)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (4)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 15 (32)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 6 (6) — Scattered macular rash across back; mild skin rash left mid lower back; Rash on shins/calves; Blisters Rt thigh/hip area; generalized erythema/edema; ulceration sacral region. ulceration right labia majora; skin breakdown under flange of j-tube
Flushing (Vascular disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (5)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Glucose intolerance (Metabolism and nutrition disorders) | 17 (23)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-05-05): https://cdn.clinicaltrials.gov/large-docs/90/NCT03064490/Prot_SAP_000.pdf
  • Informed Consent Form (2022-07-20): https://cdn.clinicaltrials.gov/large-docs/90/NCT03064490/ICF_001.pdf